CLINICAL TRIAL: NCT02365532
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Oral GS-6615 on Dofetilide-Induced QT Prolongation, Safety, and Tolerability in Healthy Subjects
Brief Title: Effect of Oral GS-6615 on Dofetilide-Induced QT Prolongation, Safety, and Tolerability in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-372-1666
Record Dates: First submitted 2015-02-13; First posted 2015-02-19 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Long QT Syndrome
Keywords: drug-induced long QT syndrome; DILQTS; prolonged QT
MeSH Terms: conditions — Long QT Syndrome | interventions — eleclazine; dofetilide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo to match GS-6615 (Placebo Comparator): Placebo to match GS-6615 + dofetilide or placebo to match dofetilide twice daily
  Interventions: Drug: Placebo to match GS-6615; Drug: Placebo to match dofetilide; Drug: Dofetilide
- GS-6615 (Experimental): GS-6615 or placebo to match GS-6615 + dofetilide or placebo to match dofetilide twice daily
  Interventions: Drug: GS-6615; Drug: Placebo to match GS-6615; Drug: Placebo to match dofetilide; Drug: Dofetilide

INTERVENTIONS:
Drug: GS-6615 — GS-6615 tablets administered orally
  Arms: GS-6615
Drug: Placebo to match GS-6615 — Placebo to match GS-6615 tablets administered orally
Drug: Placebo to match dofetilide — Placebo to match dofetilide capsules administered orally
Drug: Dofetilide — Dofetilide 500 μg capsules administered orally according to the current prescribing information

SUMMARY:
This study will evaluate the effect of oral GS-6615 on QTc interval in healthy adults with dofetilide-induced QTc prolongation.

ELIGIBILITY:
Inclusion Criteria:

* Must, in the opinion of the investigator, be in good health based upon medical history and physical examination, including vital signs
* Have a calculated body mass index (BMI) from 18 to 30 kg/m^2, inclusive, at study screening
* Have either a normal 12-lead electrocardiogram (ECG) or one with abnormalities that are considered clinically insignificant and which do not interfere with the ability to interpret the QT interval in the opinion of the investigator in consultation with the medical monitor

Exclusion Criteria:

* History of meningitis or encephalitis, epilepsy, seizures (known or suspected), migraines, tremors, myoclonic jerks, sleep disorder, anxiety, syncope, head injuries, or a family history of seizures
* Have any serious or active medical or psychiatric illness (including depression) which, in the opinion of the investigator, would interfere with treatment, assessment, or compliance with the protocol. This would include renal, cardiac, hematological, hepatic, pulmonary (including chronic asthma), endocrine (including diabetes), central nervous, gastrointestinal (including an ulcer), vascular, metabolic (thyroid disorders, adrenal disease), immunodeficiency disorders, active infection, or malignancy that are clinically significant or requiring treatment.
* Presence or history of cardiovascular disease, including structural heart disease, myocardial infarction (by ECG and/or clinical history), history of ventricular tachycardia or torsade de pointes, heart failure or cardiomyopathy (by clinical history and/or left ventricular ejection fraction < 40%), presence of cardiac conduction abnormalities, a family history of Long QT or Brugada Syndrome, or unexplained death in an otherwise healthy individual between the ages of 1 and 30 years
* Additional cardiovascular-specific exclusion criteria include findings on screening ECG of:

  * QTcF interval > 430 msec
  * PR interval > 220 msec
  * QRS duration > 110 msec
  * Second- or third-degree atrioventricular block
  * Complete left or right bundle branch block or incomplete right bundle branch block
  * Resting heart rate < 40 or > 100 beats per minute (bpm)
  * Pathological Q waves (defined as Q wave > 40 msec)
  * Ventricular pre-excitation
  * More than 2 ectopic beats
* Syncope, palpitations, or unexplained dizziness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in daytime QT interval corrected for heart rate using the Fridericia formula (QTcF) | Up to 6 days
Pharmacokinetic (PK) profiles of GS-6615 and dofetilide | Predose and postdose on Days -2 through Day 4
  This endpoint will measure the plasma PK profiles of GS-6615 and dofetilide. PK parameters that will be measured include Cmax, Tmax, AUC_0-24, and AUC_0-tlast.

SECONDARY OUTCOMES:
Incidence of adverse events, clinical laboratory test results, vital sign measurements, and electrocardiogram (ECG) data | Up to 6 days
  This endpoint will measure the safety and tolerability profile of GS-6615.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly B Patel, MD, Study Director — Gilead Sciences
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States